CLINICAL TRIAL: NCT06548815
Title: A Single-center, Single-administration, Randomized, Placebo-controlled, Dose-escalation Trial Evaluated the Safety, Tolerability, PK, and PD Parameters of GZR4 in Healthy Male Adult Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single-dose GZR4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GL-GZR-CH1004
Record Dates: First submitted 2024-08-05; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Diabetes
Keywords: GZR4; PK
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GZR4 (Experimental): s.c, single dose
  Interventions: Drug: GZR4
- Placebo (Placebo Comparator): s.c, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GZR4 — Ascending single doses - 4 dose levels.
  Arms: GZR4
Drug: Placebo — Ascending single doses - 4 dose levels.
  Arms: Placebo

SUMMARY:
This trial is conducted in China. The aim of this trial is to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of single-dose GZR4.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy male adult subjects aged 18-45 years old
* Body mass index [BMI between 19.0-24.0 kg/m2
* Hemoglobin A1c (HbA1c)≤6%

Exclusion Criteria:

* Abnormalities that were assessed by the investigators to be clinically significant at screening included vital signs, physical examination, laboratory testing, anteroposterior and lateral chest radiography, and 12-lead ECG
* Known severe allergies (e.g., allergy to more than 3 allergens, allergic asthma affecting the lower respiratory tract, allergy requiring glucocorticoid treatment) or known allergic history to the ingredients of the investigational drug used in this study
* Participants had donated blood ≥ 200 mL within 6 months before screening, or had donated blood components, or had a total blood loss of ≥ 200 mL due to any reason, or history of blood transfusion or use of blood products
* Human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or treponema pallidum antibody positive
* Participated in other clinical trials and used investigational drugs or medical devices within 3 months before screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Incidence of TEAE | Baseline to Day29

SECONDARY OUTCOMES:
GIRmax | Day2-Day3
Tmax,GIR | Day2-Day3
AUCGIR | Day2-Day3/Day7-Day8
Cmax | Baseline to Day29
Tmax,GZR4 | Baseline to Day29
T1/2 | Baseline to Day29
AUC0-inf | Baseline to Day29
AUC0-last | Baseline to Day29

CONTACTS AND LOCATIONS:
Locations (1):
- Gan & Lee Pharmaceuticals Co., Ltd, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No